CLINICAL TRIAL: NCT06549907
Title: A Biomarker Exploratory Study of Efficacy and Prognosis of Dual Blockade of PD1/PDL1 and CTLA4 in Combination of Anti-angiogenic Treatment in MSS Metastatic Colorectal Cancers and MSI Solid Tumors Refractory to PD1/PDL1 Antibody Monotherapy
Brief Title: A Biomarker Exploratory Study of Dual Blockade of PD1/PDL1 and CTLA4 and Anti-angiogenic Therapy
Status: Recruiting | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CGOG-EXPLORE-03
Record Dates: First submitted 2023-11-10; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: MSS Metastatic Colorectal Cancers; MSI Solid Tumors Refractory to PD1/PDL1 Antibody Monotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Exploratory group: Patients treated with dual blockade of PD1/PDL1 and CTLA4 in combination of anti-angiogenic treatment
  Interventions: Other: Multi-omics testing; Other: MRI

INTERVENTIONS:
Other: Multi-omics testing — Samples include tissue, blood, urine and stool, and multi-omics approaches include single-cell sequencing, spatial transcriptome sequencing, macro transcriptome sequencing, whole exome sequencing, microproteomics, immunohistochemistry, and multiplex fluorescence immunohistochemistry.
Other: MRI — MRI will be conducted to investigate image characteristics during treatment

SUMMARY:
This study is a single-center prospective exploratory research, aiming to identify clinical characteristics and biomarkers associated with the therapeutic effects of dual PD1/PDL1 and CTLA4 blockade plus anti-angiogenic therapy and investigate MR image characteristics during treatment in patients with MSS metastatic colorectal cancer and MSI solid tumors resistant to PD-1/PD-L1 antibody monotherapy.

DETAILED DESCRIPTION:
This study is a single-center prospective exploratory research. Patients with MSS metastatic colorectal cancer and MSI solid tumors resistant to PD-1/PD-L1 antibody monotherapy who are treated with dual PD1/PDL1 and CTLA4 blockade combined with anti-angiogenic therapy in the Department of Gastrointestinal Oncology of Peking University Cancer Hospital will be enrolled. Their clinical-pathological features and specimens will be collected at baseline, at each tumor assessment point, and at disease progression.

This study aims to identify clinical characteristics and biomarkers associated with the therapeutic effects through multi-omics approaches, and to investigate MR image characteristics during treatment. Samples include tissue, blood, urine and stool, and multi-omics approaches include single-cell sequencing, spatial transcriptome sequencing, macro transcriptome sequencing, whole exome sequencing, microproteomics, immunohistochemistry, and multiplex fluorescence immunohistochemistry.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed MSS metastatic colorectal cancers or MSI solid tumors refractory to PD1/PDL1 antibody monotherapy
* Receiving dual blockade of PD1/PDL1 and CTLA4 in combination of anti-angiogenic treatment with or without other therapies

Exclusion Criteria:

●Having malignancies in non-gastrointestinal system that have not been cured (Lynch syndrome not included)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with MSS metastatic colorectal cancer and MSI solid tumors resistant to PD-1/PD-L1 antibody monotherapy who are treated with dual PD1/PDL1 and CTLA4 blockade plus anti-angiogenic therapy
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Baseline proportion and location of different immune cell subsets associated with efficacy | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Proportion and location of different immune cell subsets will be assessed by single-cell sequencing, spatial transcriptome sequencing, immunohistochemistry, and multiplex fluorescence immunohistochemistry using pre-treatment samples.
Baseline tumor gene alterations associated with efficacy | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Baseline tumor gene alterations will be assessed by whole exome sequencing using pre-treatment tissue or blood samples
Baseline clinical characteristics associated with efficacy | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Baseline clinical characteristics include age of onset, gender, family history, pathological type of tumor, primary tumor site, metastatic site, tumor size, and previous treatment.
Baseline tumor-associated proteins associated with efficacy | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Tumor-associated proteins will be assessed by microproteomics using pre-treatment blood or urine samples.
Baseline intestinal flora associated with efficacy | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Intestinal flora will be assessed by macro transcriptome sequencing using pre-treatment stool samples.

SECONDARY OUTCOMES:
Early changes (within 8 weeks) of proportion and location of different immune cell subsets after treatment associated with efficacy | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Proportion and location of different immune cell subsets will be assessed by single-cell sequencing, spatial transcriptome sequencing, immunohistochemistry, and multiplex fluorescence immunohistochemistry using pre-and post-treatment samples.
Early changes (within 8 weeks) of tumor gene alterations after treatment | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Baseline tumor gene alterations will be assessed by whole exome sequencing using pre-and post-treatment tissue or blood samples.
Early changes (within 8 weeks) of tumor-associated proteins after treatment associated with efficacy | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Tumor-associated proteins will be assessed by microproteomics using pre-and post treatment blood or urine samples.
Early changes (within 8 weeks) of intestinal flora after treatment associated with efficacy | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Intestinal flora will be assessed by macro transcriptome sequencing using pre- and post-treatment stool samples.
Longitudinal on-treatment changes of proportion and location of different immune cell subsets at baseline, tumor shrinkage and progression | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Proportion and location of different immune cell subsets will be assessed by single-cell sequencing, spatial transcriptome sequencing, immunohistochemistry, and multiplex fluorescence immunohistochemistry using pre-and post-treatment samples.
MR image characteristics | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  MR image characteristics at baseline and their changes when tumor responded or progressed

CONTACTS AND LOCATIONS:
Overall Officials: Jian Li, Study Director — Peking University Cancer Hospital & Institute
Locations (1):
- Jian Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No